CLINICAL TRIAL: NCT05224531
Title: A Phase 2, Prospective, Randomized, Open-label, Blinded Endpoint, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy of 3 Doses of CS1 in Subjects With Pulmonary Arterial Hypertension
Brief Title: Effect of CS1 in Subjects With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cereno Scientific AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS1-003
Record Dates: First submitted 2022-01-17; First posted 2022-02-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; CARDIOMEMS
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded Endpoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CS1 480 mg dose group (Experimental): 480 mg of CS1, twice daily administration with 1/3 of the dose in the morning and 2/3 in the evening.
  Interventions: Drug: CS1 Administration
- CS1 960 mg dose group (Experimental): 960 mg of CS1, twice daily administration with 1/3 of the dose in the morning and 2/3 in the evening.
  Interventions: Drug: CS1 Administration
- CS1 1920 mg dose group (Experimental): 1920 mg of CS1, twice daily administration with 1/3 of the dose in the morning and 2/3 in the evening.
  Interventions: Drug: CS1 Administration

INTERVENTIONS:
Drug: CS1 Administration — CS1 delayed-release capsules will be supplied with 160 mg active pharmaceutical ingredient (sodium valproate) per capsule. Three dose levels that will be evaluated in this study; study drug will be administered as uneven, divided doses twice daily in the morning and in the evening (1/3 of the daily dose is to be administered between 7 and 9 am; 2/3 of the daily dose is to be administered between 7 and 9 pm).

SUMMARY:
This is a Phase 2, parallel group study to evaluate the safety, tolerability, PK, and exploratory efficacy of 3 doses of CS1 in the treatment of PAH using the CardioMEMS HF System to obtain repeated measurements of PAP and other hemodynamic parameters.

Elegible subjects will have a RHC to implant the CardioMEMS pulmonary artery (PA) Sensor followed by a Baseline Period for the subject to become familiar with the system, its measurements, how to send the data, and establish Baseline PA pressure. Alternately, the subject may already have the CardioMEMS HF System and is willing to have the system recalibrated in conjunction with RHC. Thereafter, the subject will be randomly assigned to 1 of 3 total daily doses of CS1 1:1:1; there will be 10 subjects assigned to each dose level. Subjects will receive study drug treatment for 12 weeks. During the study, mPAP and other hemodynamic parameters from CardioMEMS PA Sensor will be measured and data captured once daily in the morning before the subject gets out of bed.

The data will be transferred electronically to a repository. The analysis will look at the area under the curve (AUC) of mPAP and the doses will be compared to each other regarding change from Baseline. In addition to the CardioMEMS HF System measurements, the subjects will be followed for mortality and morbidity, important biomarkers as well as subjective, functional, and structural parameters of importance for PAH, for the duration of the study.

Subjects will be enrolled for up to 22 weeks: a Screening Period of up to 2 weeks prior to the start of the Baseline Period, a Baseline Period of up to 6 weeks prior to Randomization, a Treatment Period of 12 weeks, and a Follow-up Period of 2 weeks.

The primary objective of the study is to obtain safety and tolerability data.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for inclusion in the study if they meet all of the following criteria:

1. Subject must be willing and able to sign a written informed consent prior to any study-related procedures and able to understand and follow instructions; return to the study unit for specified study visits; and able to participate in the study for the entire period.
2. Subject is male or female, aged 18 to 80 years.
3. Subject must have a body mass index (BMI) 18 to 40 kg/m2 at Screening. If BMI is >35 kg/m2, subject chest circumference should be <65 inches (165 cm).
4. Subject with PAH belonging to 1 of the following subgroups of NICE Clinical Classification of PAH category:

   1. Idiopathic PAH.
   2. Heritable PAH.
   3. Drug or toxin-induced (anorexigen or methamphetamine use).
   4. PAH associated with connective tissue disease.
5. Subject with PAH who are symptomatic and have reduced exercise capacity due primarily to their PAH diagnosis, having been assessed by qualified individual, ie, physician, physician assistant, or nurse practitioner, to be in NYHA/WHO functional class II or III and having an RRS 2.0 of 6 to 10.
6. PAH therapy at stable doses of standard-of-care therapies for at least 90 days prior to screening.
7. Subject has most recent (within the last 36 months) hemodynamic assessment of PAH by RHC demonstrating a persistent resting mPAP ≥25 mm Hg and resting mean pulmonary vascular resistance (PVR) ≥5 Wood Units with Pulmonary Capillary Wedge Pressure ≤15 mmHg.
8. Subject is willing to undergo CardioMEMS PA Sensor implantation and RHC prior to randomization or has had the CardioMEMS PA Sensor implanted previously.
9. Subject has a 6-minute walk distance (6MWD) ≥150 meters (m) and <550 m at Screening.
10. Female subject of childbearing potential must be willing and able to practice effective contraception during the study and continuing contraception for 30 days after their last dose of study drug. A female subject of non-childbearing potential is defined as being surgically sterilized by bilateral tubal ligation, bilateral oophorectomy, or hysterectomy. A female subject 45 to 60 years of age, who is post-menopausal for at least 1 year, and has a follicle-stimulating hormone level confirmation indicating post menopausal status will be considered of non-childbearing potential. A female subject >60 years of age is considered post menopausal and of non childbearing potential.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Subject has pulmonary hypertension category 2 to 5.
2. Subject has adult congenital heart disease (ACHD).
3. Subject has concomitant medical or psychiatric disorder, condition, history, or any other condition that in the opinion of the Investigator would either put the subject at risk or impair the subject's ability to participate in or complete the requirements of the study or confound the objectives of the study.
4. Subject has a concomitant medical disorder that is expected to limit the subject's life-expectancy to ≤1 year.
5. Subject has RRS 2.0 score of ≤5 or ≥11.
6. Subject has heart fai
7. lure with preserved ejection fraction defined as those with >50% ejection fraction (with signs and symptoms of heart failure) or left atrial volume (LAV) >34 mL/ m2.
8. Subject is not able to have CardioMEMS PA Sensor implanted due to:

   1. An active, ongoing infection defined as being febrile, an elevated white blood cell count, on intravenous antibiotics, and/or positive cultures (blood, sputum, or urine).
   2. History of current or recurrent (≥2 episodes within 5 years prior to consent) pulmonary emboli and/or deep vein thromboses.
   3. Cannot tolerate RHC.
   4. PA branch inner diameter <7 mm in a descending branch within the left or right lower lung lobe (target implant vessel).
   5. Unable to take dual antiplatelet or anticoagulation therapy for 1 month after CardioMEMS PA Sensor implantation.
9. Subject is likely to undergo lung transplantation within the next 6 months.
10. Subject has untreated, moderate to severe obstructive sleep apnea.
11. Subject has evidence of significant chronic thromboembolic disorder as determined by the Investigator or recent pulmonary embolism within 6 months prior to Screening (see also exclusion criterium 7b).
12. Subject has uncontrolled hypertension (˃160/100 mmHg, confirmed by duplicate seated readings) at 2 or more historical visits within 3 months prior to Screening.
13. Subject has sustained systolic blood pressure <95 mmHg and/or diastolic blood pressure <50 mmHg (confirmed by duplicate seated readings) on at least 3 consecutive occasions (self monitored or office) prior to or at Screening, or overt symptomatic hypotension.
14. Subject has sustained resting heart rate >120 beats per minute (confirmed by duplicate assessments of office vital signs) or consecutive electrocardiogram (ECG) assessments on at least 3 consecutive occasions prior to or at Screening.
15. Subject has a history of a bleeding disorder.
16. Subject has thrombocytopenia: platelets <150,000/mm3.
17. Subject has known porphyria, mitochondrial, or urea cycle disease.
18. Subject has a history of chronic pancreatic disease.
19. Subject is a pregnant or lactating female.
20. Subject has a positive result from serology testing at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV); but if the subject has a historical diagnosis (prior to Screening) of being positive for HIV, HBsAg, or HCV, must be clinically stable and if on therapy, be on stable therapy for at least 3 months prior to Screening. A subject should not have active coronavirus disease 19 (COVID-19); however, those with previous COVID 19 are permitted.
21. Subject has participated in another investigational drug study within 30 days prior to Screening or is participating in a non medication study which, in the opinion of the Investigator, would interfere with the study compliance or outcome assessments.
22. Subject is on regular treatment with sodium valproate/valproic acid (VPA), other anti-epilepsy drugs, or other prohibited medications that cannot be discontinued at the Screening Visit (V1).
23. Subject is on regular anticoagulation or on dual antiplatelet therapy (DAPT) that cannot be discontinued at the Screening Visit (V1); however, during the Baseline Period following CardioMEMS PA Sensor implantation, DAPT is allowed according to clinical practice for up to 4 weeks. A low daily dose aspirin (<125 mg) is allowed, ie, "baby" aspirin.
24. Subject has more than mild mitral or aortic valve disease, left ventricular ejection fraction (LVEF) <50%, or left ventricular regional wall motion abnormality suggestive of active coronary artery disease on 2D-echocardiogram at Screening.
25. Subject has a forced expiratory volume in 1 second (FEV1)/forced vital capacity <70% (absolute), FEV1 ≤50% or total lung capacity (TLC) <70% predicted on pulmonary function testing (PFT); for potential subjects with TLC 60 to 69% predicted, non contrasted computerized tomography (CT) scan must be performed to exclude subjects with more than mild interstitial lung disease. PFTs should have been obtained within 3 years prior to Screening.
26. Subject has clinically significant renal dysfunction as measured by the estimated Glomerular Filtration Rate (eGFR) of <30 mL/min/1.73m2 as calculated by Modification of Diet in Renal Disease (MDRD) at Screening.
27. Subject has significant liver dysfunction as measured by any one of the following at Screening (including subjects with acute or chronic hepatitis as well as subjects with own or family history of serious hepatitis, especially drug related):

    1. Alanine aminotransferase (ALT) >2.0 × upper limit of normal (ULN).
    2. Aspartate aminotransferase (AST) >2.0 × ULN.
    3. Serum bilirubin ≥1.6 mg/dL or >2.0 × ULN.
28. Subject has a known history of substance abuse including alcohol abuse within the 1 year prior to Screening that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study.
29. Subjects with any major surgical procedure or trauma within 30 days prior to Screening or planned surgical procedure during the study period.
30. Subject with any inpatient hospitalization (defined as >23 hours) within 30 days prior to Screening.
31. Subject enrolled within 90 days prior to Screening or plans to enroll during the study into a cardiopulmonary rehabilitation program.
32. Subject has known hypersensitivity to study drug or any of the excipients of the drug formulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Patient reported adverse events | 6 months
  Safety and tolerability of 3 doses of CS1

CONTACTS AND LOCATIONS:
Locations (1):
- Fredrik Frick, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided